CLINICAL TRIAL: NCT03029611
Title: A Phase II Study of Concurrent IGFBP-2 Vaccination and Neoadjuvant Chemotherapy to Increase the Rate of Pathologic Complete Response at the Time of Cytoreductive Surgery
Brief Title: IGFBP-2 Vaccine and Combination Chemotherapy in Treating Patients With Stage III-IV Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Undergoing Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to lack of funding
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary (Nora) Disis, Professor, Department of Medicine, Division of Oncology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9760; NCI-2017-00034 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1717017 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2017-01-10; First posted 2017-01-24 (Estimated); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Stage III Fallopian Tube Cancer; Stage III Ovarian Cancer; Stage III Primary Peritoneal Cancer; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; Gynecologic Surgical Procedures; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, IGFBP-2 vaccine) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour followed by IGFBP-2 vaccine ID 2 weeks later. Treatment repeats every 3 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. After completion of 3 cycles, patients then undergo cytoreductive surgery.
  Interventions: Drug: Carboplatin; Procedure: Gynecological Surgical Procedure; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: pUMVC3-hIGFBP-2 Multi-Epitope Plasmid DNA Vaccine

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Gynecological Surgical Procedure — Undergo cytoreductive surgery
  Other Names: gynecologic surgery; Gynecologic Surgical Procedure; gynecologic surgical procedures; gynecological surgery
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: pUMVC3-hIGFBP-2 Multi-Epitope Plasmid DNA Vaccine — Given ID

SUMMARY:
This phase II trial studies how well pUMVC3-IGFBP2 plasmid deoxyribonucleic acid (DNA) vaccine (IGFBP-2 vaccine) and combination chemotherapy work in treating patients with stage III-IV ovarian, fallopian tube, or primary peritoneal cancer undergoing surgery. IGFBP-2 is a protein found in the blood and tumor cells of most who have been diagnosed with ovarian cancer. Too much IGFBP-2 has been associated with more invasive disease. Vaccines made from DNA may help the body build an effective immune response to kill tumor cells that express IGFBP-2. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving IGFBP-2 vaccine and combination chemotherapy may work better in treating patients with stage III-IV ovarian, fallopian tube, or primary peritoneal cancer undergoing surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether the addition of an IGFBP-2 vaccine to neoadjuvant chemotherapy increases the rate of complete pathologic response (CR).

SECONDARY OBJECTIVES:

I. Determine whether the addition of an IGFBP-2 vaccine to neoadjuvant chemotherapy increases progression free survival at 12 months.

II. Determine whether the addition of an IGFBP-2 vaccine to neoadjuvant chemotherapy improves overall survival.

III. To determine whether IGFBP-2 vaccination in combination with chemotherapy increases the level of tumor infiltrating lymphocytes (TIL) in the tumor.

IV. To assess the level of IGFBP-2 type 1 helper cells (Th1) elicited with vaccination concurrent with chemotherapy.

EXPLORATORY OBJECTIVES:

I. To explore whether there is a predictive genomic signature for CR induction when IGFBP-2 vaccination is used in combination with chemotherapy.

OUTLINE:

Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 1 hour followed by IGFBP-2 vaccine intradermally (ID) 2 weeks later. Treatment repeats every 3 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. After completion of 3 cycles, patients then undergo cytoreductive surgery.

After completion of study treatment, patients are followed up at 6 months and then once a year for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed advanced stage (III/IV) ovarian cancer (ovarian/fallopian tube/peritoneal cancer) who have been recommended to receive neoadjuvant carboplatin/paclitaxel chemotherapy with subsequent cytoreductive surgery
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status score of =< 2
* Patients must have recovered from major infections and/or surgical procedures, and in the opinion of the investigator, not have any significant active concurrent medical illnesses precluding protocol treatment
* Estimated life expectancy of more than 6 months
* White blood cells (WBC) >= 3000/mm^3 within 30 days of enrollment to study
* Hemoglobin (Hgb) >= 10 g/dl within 30 days of enrollment to study
* Hematocrit (Hct) >= 28% within 30 days of enrollment to study
* Serum creatinine =< 2.0 mg/dl or creatinine clearance > 60 ml/min within 30 days of enrollment to study
* Total bilirubin =< 2.5 mg/dl within 30 days of enrollment to study
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) =< 3 times upper limit of normal (ULN) within 30 days of enrollment to study
* Blood glucose <1.5 ULN within 30 days of enrollment to study
* All patients who are having sex that can lead to pregnancy must agree to contraception for the duration of the study
* Patients must be at least 18 years of age

Exclusion Criteria:

* Patients with any of the following cardiac conditions:

  * Symptomatic restrictive cardiomyopathy
  * Unstable angina within 4 months prior to enrollment
  * New York Heart Association functional class III-IV heart failure on active treatment
  * Symptomatic pericardial effusion
* Uncontrolled diabetes
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Patients with any contraindication to receiving rhuGM-CSF based products
* Patients with any clinically significant autoimmune disease uncontrolled with treatment
* Patients who are currently receiving an anti-IGF-IR monoclonal antibody as part of their treatment regimen
* Patients who are simultaneously enrolled in any other treatment study
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Liao, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, IGFBP-2 Vaccine)
Started | 9 (We had 11 patients sign consent with 2 patients deciding not to continue to receive treatment.)
Completed | 9 (Please note that we did not fully enroll this study due to lack of funding. The complete date here relates to the last treatment administration.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 11 participants signed consent 9 participants received treatment 9 participants completed all 3 vaccines and 1 month follow-up
Arm/Group | Treatment (Chemotherapy, IGFBP-2 Vaccine)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 64 [54 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Rate of Pathologic Complete Response (CR)
Description: The tissue collected at time of cytoreductive surgery, post study treatment, was evaluated by the attending pathologist assigned to look at the tissue for viable tumor cells. The corresponding surgical pathology report was reviewed to evaluate individual pCR (absence of viable tumor cells).
Time Frame: At the time of cytoreductive surgery after receiving study treatment (vaccinations given intradermally approximately two weeks after each combination chemotherapy for 3 doses.)
Population: Review of the pathology report from cytoreductive surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, IGFBP-2 Vaccine)
Number analyzed (Participants) | 9
Participants | 0

2. Secondary Outcome: Immunohistochemistry (IHC) Staining for CD3, CD4, CD8, and CD27
Description: Will be performed and quantitated using published methods and will be correlated with surgical CR by the Man-Whitney U or one-way analysis of variance test depending on the distribution of TIL outcomes.
Time Frame: At the time of cytoreductive surgery
Population: Target enrollment was not met. Samples were collected but planned laboratory/statistical analyses were not performed due to termination of study, lack of funding, and insufficient enrollment.
Arm/Group | Treatment (Chemotherapy, IGFBP-2 Vaccine)
Number analyzed (Participants) | 0

3. Secondary Outcome: Level of IGFBP-2 Th1 Cells Elicited With Vaccine Assessed by Enzyme-linked Immunosorbent Spot Assay
Description: Will be correlated to tumor burden at definitive surgery.
Time Frame: Up to 6 months after last vaccine
Population: as for outcome 2
Arm/Group | Treatment (Chemotherapy, IGFBP-2 Vaccine)
Number analyzed (Participants) | 0

4. Secondary Outcome: Level of Tumor Infiltrating Lymphocytes (TIL) in Tumor
Description: Will be assessed by immunohistochemistry (IHC) to determine whether IGFBP-2 vaccination in combination with chemotherapy increases the level of TIL in the tumor. This was done by assessing the level of IGFBP-2 Th1 elicited by study treatment (vaccination concurrent with chemotherapy). we are looking for an increase in TIL.
Time Frame: as for outcome 1
Population: as for outcome 2
Arm/Group | Treatment (Chemotherapy, IGFBP-2 Vaccine)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Will be compared between the treatment arms. Large differences in PFS if observed between the treatment groups will be noted and described. Will be plotted by Kaplan-Meier curve, and compared to the survival data reported by Vergote et al which reported median PFS of 12 months and median OS of 30 months for patients treated with neoadjuvant chemotherapy by a log-rank test.
Time Frame: Up to 5 years
Population: Target enrollment was not met. The study was terminated. Planned statistical analysis was not performed due to termination of study, lack of funding, and insufficient enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, IGFBP-2 Vaccine)
Number analyzed (Participants) | 9
Participants
  Alive | 6
  Deceased - passed away after they left the study | 3

6. Secondary Outcome: Progression Free Survival (PFS)
Description: Large differences in PFS if observed between the treatment groups will be noted and described. Will be plotted by Kaplan-Meier curve, and compared to the survival data reported by Vergote et al which reported median PFS of 12 months and median overall survival (OS) of 30 months for patients treated with neoadjuvant chemotherapy by a log-rank test.
Time Frame: Up to 12 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, IGFBP-2 Vaccine)
Number analyzed (Participants) | 9
Participants
  PFS | 2
  Recurrence | 2
  Deceased - passed away after they left the study | 3
  Status unchanged | 2

7. Secondary Outcome: Tumor Burden
Description: Will be correlated to level of IGFBP-2 Th1 cells.
Time Frame: At the time of cytoreductive surgery
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, IGFBP-2 Vaccine)
Number analyzed (Participants) | 9
Participants
  Debulking surgery | 7
  Not evaluable | 2

8. Other Pre Specified Outcome: Predictive Signature of CR Induction When Vaccinated With an IGFBP-2 Vaccine in Combination With Neoadjuvant Chemotherapy Assessed by Whole Exome Sequencing on Vaccinated Patients' Tumors
Description: Will use the LASSO regularized regression method to generate preliminary data for a predictive signature. Will correlate mutational profiles with primary platinum sensitive, resistance and refractory outcomes, leveraging the Cancer Genome Atlas data publicly available, to determine differences induced by vaccination.
Time Frame: At the time of cytoreductive surgery
Population: as for outcome 2
Arm/Group | Treatment (Chemotherapy, IGFBP-2 Vaccine)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The Adverse Events were collected after first vaccination and through to 6 months post vaccination.
Description: We used CTCAE v4.0 for this study. The adverse events reported here include all events regardless of whether they were unrelated and related to study treatment). Please note that these tables record every adverse event for every subject regardless of severity. For example, a subject may have an injection site reaction at each of the three vaccines where another may not. Each one of these injection site reactions is recorded for that one subject.
Arm/Group | Treatment (Chemotherapy, IGFBP-2 Vaccine)
All-Cause Mortality (participants affected / at risk) | 3/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, IGFBP-2 Vaccine) (N=9)
White blood cell decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) — Unrelated to study treatment
Weight loss (Investigations) | 2 (2) — Unrelated to study treatment
Creatinine increased (Investigations) | 1 (1) — Unrelated to study treatment
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Unrelated to study treatment
Anemia (Blood and lymphatic system disorders) | 5 (6) — 4 of 6 events are unrelated to study treatment
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - leg weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - "pulled muscle" in left upper quadrant (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to study treatment
Urinary tract infection (Infections and infestations) | 2 (2) — 1 of 2 events is unrelated to study treatment
Other Infection (Infections and infestations) | 1 (1) — Unrelated to study treatment
Wound infection (Infections and infestations) | 1 (1) — Unrelated to study treatment
Palpitations (Cardiac disorders) | 2 (2) — 1 of 2 events is unrelated to study treatment
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3) — 1 of 3 events is unrelated to the study treatment
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) — Unrelated to study treatment
Nausea (Gastrointestinal disorders) | 2 (3) — 1 of 3 events is unrelated to the study treatment
Vomiting (Gastrointestinal disorders) | 2 (3) — 1 of 3 events is unrelated to the study treatment
Constipation (Gastrointestinal disorders) | 4 (5) — 2 of 5 events are unrelated to the study treatment
Abdominal distension (Gastrointestinal disorders) | 1 (1) — Unrelated to study treatment
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Unrelated to study treatment
Ascites (Gastrointestinal disorders) | 1 (1) — Unrelated to study treatment
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated to study treatment
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) — Unrelated to study treatment
Alopecia (Skin and subcutaneous tissue disorders) | 9 (12) — 1 of 12 events are unrelated to the study treatment
Fatigue (General disorders) | 2 (3)
Edema limbs (General disorders) | 1 (1) — Unrelated to study treatment
Non-cardiac chest pain (General disorders) | 1 (1) — Unrelated to study treatment
Pain (General disorders) | 5 (6) — 5 of 6 events are unrelated to the study drug
Injection site reaction (General disorders) | 4 (4)
Flushing (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) — Unrelated to study treatment
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) — Unrelated to study treatment
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) — Unrelated to study treatment
Cystitis noninfective (Renal and urinary disorders) | 1 (1) — Unrelated to study treatment
Hematuria (Renal and urinary disorders) | 1 (1) — Unrelated to study treatment
Acute kidney injury (Renal and urinary disorders) | 1 (1) — Unrelated to study treatment
Other - paracentisis (Surgical and medical procedures) | 4 (4) — Unrelated to study treatment
Other - IVC filter placed due to clots (Surgical and medical procedures) | 1 (1) — Unrelated to study treatment
Other - thoracentesis x 2 due to pleural effusion. Hospitalized (Surgical and medical procedures) | 1 (1) — Unrelated to study treatment
Other - ex-lap, RSO, omentectomy, appendectomy, tumor debulking (Surgical and medical procedures) | 1 (1) — Unrelated to study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03029611/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03029611/ICF_002.pdf